CLINICAL TRIAL: NCT04994028
Title: Effectiveness of Volume Spirometry and Deep Breathing Exercise for Dyspnea During Third Trimester of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0301 Uzma Batool
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Dyspnea; Pregnancy Related
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Conventional treatment that include behavioral and life style modification and dyspnea prevention education
  Interventions: Other: Conventional treatment
- conventional treatment with volume Spirometry and deep breathing (Experimental): Conventional treatment along with volume Spirometry and deep breathing exercise
  Interventions: Other: conventional treatment with volume Spirometry and deep breathing

INTERVENTIONS:
Other: Conventional treatment — Behavioral and life style modification and dyspnea prevention education i.e. Sitting: Sit upright with back against chair, feet wide apart, leaning forward with arms on bedside table or on knees. Standing: Lean back against wall with feet slightly apart with head and shoulder relaxed. In Bed: Elevate head of the bed, support and elevate arms with pillow. Stairs: Lean forward with on banister when climbing stairs.
  Arms: Conventional treatment
Other: conventional treatment with volume Spirometry and deep breathing — Group B or interventional group was received conventional treatment along with volume Spirometry and deep breathing exercise, total 5 breaths with 3sec inhalational breath hold for each breath at one session per day for volume Spirometry and for deep breathing exercise 10 times with breath hold 2sec at every session for 5 minutes 3 times per week for total duration of two weeks.
  Arms: conventional treatment with volume Spirometry and deep breathing

SUMMARY:
During pregnancy women undergoes anatomical, mechanical and physiological changes to meet the demand of growing fetus. Dyspnea is a common complaint in pregnancy related to change in respiratory centre threshold and sensitivity. Pregnant women who engaged in regular exercise have less pregnancy induced discomforts like dyspnea and leg cramps than who did not engage in exercise. During pregnancy women undergoes anatomical, mechanical and physiological changes to meet the demand of growing fetus. Purpose of this study was to evaluate the efficacy of volume Spirometry and breathing exercise on dyspnea in third trimester of pregnancy. Rationale of the study was to find the effects of volume Spirometry and breathing exercise on dyspnea with focus on method of deep breathing exercise and volume Spirometry and outcomes. Significance of this study was to improve functional capacity and quality of life in pregnancy induced dyspnea. Subjects were randomly allocated to either two groups both groups received baseline treatment while interventional group received volume Spirometry and deep breathing exercise. Estimated sample size of 48 divided into 24 in either group by randomization. Modified Borg scale and visual analog scale were used to collect the findings. Non-parametric tests were used and analyzed by using spss22.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-30
* Primigravida and multigravida with 3rd trimester
* Singleton and twin pregnancy

Exclusion Criteria:

* Cardiac and respiratory disorders
* Smoker
* Obesity
* Any type of allergy
* Autoimmune disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Modified dyspnea Borg scale | 2nd week
  Modified Borg Dyspnea Scale is most commonly used to assess symptoms of breathlessness. It has a range from 0 to 10 (with 0 being no exertion and 10 being maximum effort).
Modified Medical Research Council Dyspnea Scale (mMRC) | 2nd week
  Questionnaire that consist of 5 statements about breathlessness. Grade0, get breathlessness only at strenuous exercise. Grade1, got breathlessness when hurrying on level ground. Grade2, walk slower than the people of my age on the level. Grade3, stop for breath after few minutes of walk on the level. Grade4, too breathlessness to leave the house when dressing or undressing.
London chest activity of Daily Living questionnaire (LCADL) | 2nd week
  It consist of four domains Selfcare, domestic activities, physical activities and leisure activities.
  Selfcare, domestic, physical and leisure activities contains 4, 6, 2 and 3 items respectively. Each item is graded by numbers 0-5, 0 mean little or no dyspnea and 5 mean worst dyspnea.gy

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Teaching Hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolomanska D, Zarawski M, Mazur-Bialy A. Physical Activity and Depressive Disorders in Pregnant Women-A Systematic Review. Medicina (Kaunas). 2019 May 26;55(5):212. doi: 10.3390/medicina55050212. PMID 31130705
- [Background] Jensen D, Ofir D, O'Donnell DE. Effects of pregnancy, obesity and aging on the intensity of perceived breathlessness during exercise in healthy humans. Respir Physiol Neurobiol. 2009 May 30;167(1):87-100. doi: 10.1016/j.resp.2009.01.011. Epub 2009 Feb 7. PMID 19450766
- [Background] Bidad K, Heidarnazhad H, Pourpak Z, Ramazanzadeh F, Zendehdel N, Moin M. Frequency of asthma as the cause of dyspnea in pregnancy. Int J Gynaecol Obstet. 2010 Nov;111(2):140-3. doi: 10.1016/j.ijgo.2010.05.024. Epub 2010 Aug 12. PMID 20708180
- [Background] Chiron B, Laffon M, Ferrandiere M, Pittet JF, Marret H, Mercier C. Standard preoxygenation technique versus two rapid techniques in pregnant patients. Int J Obstet Anesth. 2004 Jan;13(1):11-4. doi: 10.1016/S0959-289X(03)00095-5. PMID 15321433
- [Background] Nurcahyani AS, Runjati R, Nugraheni SA. Giving Belly Breathing Technique and Positive Affirmation of Stress and Cortisol Hormone Levels in Third Trimester Pregnant Women. 2020. 77. Fiskin G, Sahin NH. Effect of diaphragmatic breathing exercise on psychological parameters in gestational diabetes: A randomised controlled trial. European Journal of Integrative Medicine. 2018;23:50-6
- [Background] Armstrong CO. Post-op incentive spirometry: Why, when, & how. Nursing. 2017 Jun;47(6):54-57. doi: 10.1097/01.NURSE.0000516223.16649.02. No abstract available. PMID 28538354